CLINICAL TRIAL: NCT01188005
Title: Inflammatory Mediators in Obstructive Sleep Apnoea Syndrome; Mechanisms of Production and the Effect of Long Term Antioxidants Administration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Associate Professor Theodoros Vassilakopoulos, University of Athens Medical School
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 439
Record Dates: First submitted 2010-08-20; First posted 2010-08-25 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2010-08

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: OSAS; Sleep Apnoea; IL6; TNFα; Oxidative Stress; Antioxidants
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Vitamin A; Ascorbic Acid; Vitamin E; Allopurinol; Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OSAS patients (Experimental): This arm includes the OSAS diagnosed cohort that has been planned to undergo four polysomnographic studies. One standard, one with oxygen supplementation, one with n-CPAP device and one post antioxidants administration
  Interventions: Device: n-CPAP; Device: Oxygen supplementation; Drug: Vitamin A, Vitamin C, Vitamin E, Allopurinol, N-Acetylcysteine
- Control Group (No Intervention): This group is scheduled to undergo a plain polysomnographic study, whilst plasma cytokine levels will be measured. It will comprise of healthy, non-OSAS volunteers.

INTERVENTIONS:
Device: n-CPAP — administration of continuous positive airway pressure through a nasal device
  Arms: OSAS patients
Device: Oxygen supplementation — Oxygen supplementation (3L) through nasal spectacles
  Arms: OSAS patients
Drug: Vitamin A, Vitamin C, Vitamin E, Allopurinol, N-Acetylcysteine — Vitamin A 50,000 IU, Vitamin C 1000 mg , Vitamin E 200 mg, Allopurinol 600 mg, N-Acetylcysteine 2 g. Duration is set for 60 days
  Arms: OSAS patients

SUMMARY:
Obstructive Sleep Apnea Syndrome (OSAS) is associated with elevated plasma levels of IL-6 and TNF-α, which cannot be accounted for by obesity (Vgontzas et al Sleep Med Rev 2005;9:211-24, Ciftci et al Cytokine 2004;28:87-91].

Obstructive apneas-hypopneas are accompanied by strenuous diaphragmatic contractions before the ensuing arousals and re-establishment of airway patency. We have shown that strenuous diaphragmatic contractions induced by resistive loading lead to elevated plasma levels of IL-6, TNF-α, and IL-1β (Vassi-lakopoulos et al AJRCCM 2002;166:1572-8) with concomitant up-regulation of the cytokines within the diaphragmatic myofibers (Vassilakopoulos et al AJRCCM 2004;170:154-61).

OSAS patients exhibit frequent episodes of hypoxemia during the night. Loaded breathing is a form exercise for the respiratory muscles, and both acute and chronic hypoxia lead to an augmented plasma IL-6 response to exercise compared to normoxia (Lundby et al Eur J Appl Physiol 2004;91:88-93).

In OSAS, monocytes have oxidative stress (Dyugovskaya et al AJRCCM 2002;165:934-9) and produce more cytokines (TNF-α) in vitro (Minoguchi et al Chest 204;126:1473-9).

Hypothesis #1: plasma levels of IL-6 and TNF-α are increased during the night in OSAS patients secondary to the intermittent strenuous diaphragmatic contractions and the episodes of hypoxia-reoxygenation associated with the obstructive apneas-hypopneas.

Hypothesis #2: monocytes from sleep apnea patients, exhibit augmented intracellular expression of IL-6 and TNF-α during the night.

Hypothesis #3: Oxidative stress is a stimulus for cytokine upregulation in OSAS.

ELIGIBILITY:
Inclusion Criteria:

* Obstructive Sleep Apnea Syndrome diagnosis

Exclusion Criteria:

* narcolepsy or idiopathic hypersomnia
* chronic obstructive disease,
* neuromuscular or endocrinological disease,
* autoimmune systemic disease,
* psychological disorders,
* use of non steroids antinflammatory drugs,
* use of cortisone drugs,
* recent or concomitant systemic infections
* upper or lower airway infections

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-08; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
IL-6 Area under the curve | three months
  The primary outcome measure ( IL-6 Area under the curve) is evaluated at the end of each polysonographic study. We anticipate each subject to have completed all three sudies within one month and receive the antioxidant supplementation for an additional 60 day period. In total three months

SECONDARY OUTCOMES:
TNF-a area under the curve | three months
  The secondary outcome measure ( TNF-a Area under the curve) is evaluated at the end of each polysonographic study. we anticipate each subject to have completed all three sudies within one month and receive the antioxidant supplementation for an additional 60 day period. In total three months

CONTACTS AND LOCATIONS:
Overall Officials: Theodoros Vassilakopoulos, MD, PhD, Principal Investigator — Associate Professor in Critical Care, University of Athens
Locations (1):
- Department of Critical Care Evangelismos General Hospital, Athens, Attica, Greece